CLINICAL TRIAL: NCT02670031
Title: Response of the Myocardium to Hypertrophic Conditions in the Adult Population
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2603
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Left Ventricular Hypertrophy; Hypertension; Myocardial Fibrosis
Keywords: Hypertensive Heart Disease; Hypertension; Left Ventricular Hypertrophy; Myocardial Fibrosis; Cardiovascular Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from all participants.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Newly Diagnosed Hypertension: Patients will undergo the following studying procedures: electrocardiogram, echocardiogram, cardiovascular magnetic resonance imaging and 24-hr ambulatory blood pressure monitoring.
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Echocardiogram; Other: Electrocardiogram; Device: Ambulatory Blood Pressure Monitoring; Other: Retinal Photography (Optional)
- Well-Controlled Hypertension: Patients will undergo the following studying procedures: electrocardiogram, echocardiogram, cardiovascular magnetic resonance imaging and 24-hr ambulatory blood pressure monitoring.
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Echocardiogram; Other: Electrocardiogram; Device: Ambulatory Blood Pressure Monitoring; Other: Retinal Photography (Optional)
- Resistant Essential Hypertension: Patients will undergo the following studying procedures: electrocardiogram, echocardiogram, cardiovascular magnetic resonance imaging and 24-hr ambulatory blood pressure monitoring.
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Echocardiogram; Other: Electrocardiogram; Device: Ambulatory Blood Pressure Monitoring; Other: Retinal Photography (Optional)

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance — For the evaluation of left ventricular volumes, function and mass. This is also for the assessment of myocardial fibrosis based on delayed enhancement imaging technique.
Other: Echocardiogram — For the assessment of diastolic and systolic function as well as valvular and cardiac function. Ventricular-arterial coupling will also be performed.
Other: Electrocardiogram — To examine specific function of the heart.
Device: Ambulatory Blood Pressure Monitoring — A 24-hour test.
Other: Retinal Photography (Optional) — The test studies the structure and function of the eye vessels. It involves using eye drops to dilate the pupils, allowing the retinal photographer to have a better view of the back of the eye.

SUMMARY:
Hypertension and aortic stenosis are the two leading conditions that cause thickening of the heart muscles (left ventricular hypertrophy). Left ventricular hypertrophy is initially adaptive to maintain optimal heart function. Ultimately, heart failure occurs as a result of progressive muscle cell death and scarring (myocardial fibrosis). Dedicated techniques using cardiovascular magnetic resonance imaging (MRI) and novel high-sensitivity cardiac troponin blood assays are potential markers to detect myocardial fibrosis. Although hypertension-related heart disease is very common in Singapore, the significance of myocardial fibrosis is not well understood. In this study, the significance of myocardial fibrosis in 2000 patients with hypertension would be investigated. This will be the largest study using state-of-the-art MRI to examine the importance of myocardial fibrosis in hypertensive heart disease. 1000 participants, with at least 1 year follow-up, will be invited for a repeat assessment.

DETAILED DESCRIPTION:
According to the National Health Survey in 2010, more than 50% of adults between 60-69 years old in Singapore had hypertension. As the population ages and life expectancy continues to increase, an increasing incidence of hypertensive heart disease would be expected. Similar to aortic stenosis, left ventricular hypertrophy in patients with hypertension was associated with adverse cardiovascular outcome, independent of traditional risk factors including peripheral blood pressure. Unlike aortic stenosis (a condition with fixed obstruction), arterial hypertension is dynamic and with effective medical therapy, left ventricular hypertrophy can regress and outcome will improve. As such, contemporary guidelines recommend more aggressive blood pressure control in patients with hypertension and left ventricular hypertrophy. However, the correlation between arterial pressure and left ventricular mass is weak, particularly in treated individuals. Coupled with the inherent limitations of measuring peripheral blood pressure, it is clear that using arterial pressure to monitor progression or assess treatment response in patients with hypertensive heart disease is not optimal.

Without timely and appropriate therapies, left ventricular hypertrophy will become progressively maladaptive and ultimately the heart fails. Whilst heart failure is more commonly known by the signs and symptoms related to impaired systolic ejection fraction, heart failure with preserved ejection fraction is an increasingly recognized complex entity characterized by signs and symptoms of heart failure in the presence of preserved ejection fraction. To date, therapies that improve outcomes in heart failure with reduced ejection fraction have not shown similar benefits in patients with heart failure and preserved ejection fraction. There is no single explanation for these negative findings, but one potential reason may relate to the heterogeneity of patients recruited into these trials, and thus supporting a more targeted approach to specific phenotypes rather than a standard treatment strategy for all patients.

Therefore, a focus on the transition from compensatory left ventricular hypertrophy to ventricular decompensation is crucial not only in furthering our understanding of the pathophysiology of hypertensive heart disease, but also instrumental in designing future trials. Small studies had reported replacement myocardial fibrosis in patients with hypertension. But these studies were small and unable to establish determinants associated with myocardial fibrosis. Unlike the increasing evidence of myocardial fibrosis in aortic stenosis, the prognosis associated with myocardial fibrosis in patients with hypertension is currently not known. Although there is promising data suggesting regression in myocardial fibrosis with certain antihypertensive therapies, the effects of myocardial fibrosis regression on long-term outcome is not known. As discussed earlier, other than relying on peripheral blood pressure, there are no biomarkers to monitor response of antihypertensive therapy on regression of left ventricular mass and myocardial fibrosis.

Our investigators would establish a paradigm to demonstrate the significance of myocardial fibrosis in hypertensive heart disease; and examine other biomarkers associated with myocardial fibrosis and myocyte death that have high potential of translating into clinical application to monitor treatment response. Subsequently, the prognosis associated with myocardial fibrosis will be examined in future follow-up studies. In parallel, we will also study the effects of novel agents on the regression of left ventricular hypertrophy and myocardial fibrosis, as well as, long-term clinical outcomes in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years and over
2. Physician diagnosed essential hypertension, on at least 1 medication for blood pressure control
3. Newly diagnosed hypertension: systolic blood pressure 140mmHg or greater (diastolic blood pressure 90mmHg or greater) on at least 2 office visits (Weber 2013) and not started on any anti hypertensive medications at time of ambulatory blood pressure monitoring
4. Resistant hypertension: persistent systolic blood pressure 140mmHg or greater (diastolic blood pressure 90mmHg or greater) despite on at least 3 anti-hypertensive medications (Jennings 2013; Weber 2013)

Exclusion Criteria:

1. Known secondary hypertension: renal causes (renal artery stenosis, chronic renal failure); endocrine causes (aldosterone excess, pheochromocytoma, cushing's syndrome, hyperthyroidism); cardiac causes (coarctation of the aorta)
2. Contraindications to cardiovascular magnetic resonance: implantable devices, cerebral aneurysm clips, cochlear implants, renal impairment (GRF <30ml/min/1.73m2), claustrophobia and women who are pregnant or breast-feeding
3. Limited life expectancy
4. On-going unstable medical conditions: hypertensive crisis, acute coronary syndromes or acute heart failure
5. History of coronary artery disease, ischemic heart disease
6. History of transient ischemic attacks or cerebrovascular events
7. History of atrial fibrillation
8. History of heart failure

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from primary care clinic and outpatient clinics from the National Heart Centre Singapore. In addition, they will be recruited through posters and advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01; Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | 10 years
  Heart failure, Myocardial Infarction, Strokes and Death

CONTACTS AND LOCATIONS:
Overall Officials: Calvin WL Chin, MBBS, PhD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goh VJ, Le TT, Bryant J, Wong JI, Su B, Lee CH, Pua CJ, Sim CPY, Ang B, Aw TC, Cook SA, Chin CWL. Novel Index of Maladaptive Myocardial Remodeling in Hypertension. Circ Cardiovasc Imaging. 2017 Sep;10(9):e006840. doi: 10.1161/CIRCIMAGING.117.006840. PMID 28847911
- [Derived] Lee V, Puar T, Kui MS, Bryant JA, Han Y, Latib AB, Tay W, Kong SC, Toh DF, Boubertakh R, Lee CH, Le TT, Chin CWL. Response of the myocardium to hypertrophic conditions in the adult population (REMODEL): protocol for a prospective observational cohort study. BMJ Open. 2025 Oct 10;15(10):e100932. doi: 10.1136/bmjopen-2025-100932. PMID 41073114